CLINICAL TRIAL: NCT05051982
Title: SedLine EEG-Guided Depth of Anesthesia: Effect of Anesthetic Dosage
Brief Title: Sedline EEG Guided Depth of Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Timothy Webb, Assistant Professor of Clinical Anesthesia, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10708
Record Dates: First submitted 2021-08-23; First posted 2021-09-21 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Study Group (Experimental): Prior to the induction of anesthesia, the Sedline monitor will be placed on the patient's head to ensure the monitor is working properly. For those in the study group, the monitor will be in full view of the anesthesiologist administering the anesthetic.
  Interventions: Device: Sedline EEG in View
- Control Group (No Intervention): Prior to the induction of anesthesia, the Sedline monitor will be placed on the patient's head to ensure the monitor is working properly. For those in the control group, an apparatus will be placed over the monitor will not be in view of the anesthesiologist. The

INTERVENTIONS:
Device: Sedline EEG in View — EEG monitor (Sedline) will be in full view of the Anesthesiologist during surgery.
  Arms: Study Group

SUMMARY:
The purpose of our study is to determine if monitoring sedation (how asleep patients are under general anesthesia) using a device called a Sedline Monitor affects the amount of anesthesia patients receive.

DETAILED DESCRIPTION:
The main objective of this study is to determine if monitoring sedation using the FDA approved device, Sedline Monitor, affects the amount of anesthesia patients 65 or older receive during surgery. Reducing the anesthetic dose could result in less exposure of anesthetic medications to a high-risk patient population as well as a potential reduction in cost. Subjects will be randomized into either a control group or study group and have the Sedline Monitor placed on their head before the start of their already scheduled surgery. During the surgery, subjects in the control group will receive standard anesthesia care and the study group will receive anesthetic drug doses guided by Sedline Monitor processed EEG characteristics. When the surgery is complete, the Sedline Monitor will be removed and subject participation will be finished. The study team will also collect information about subjects from their medical records and use it for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a scheduled surgery (laparotomy, hepatobiliary surgery, gynecologic surgery, and/or urologic surgery procedures) at Indiana University Health University Hospital that is expected to have at least a 3 day post-operative hospital stay.
* ASA class 1, 2, 3, or 4.
* Age 65 years or older.
* Male or Female
* Surgical procedure requiring general anesthesia.

Exclusion Criteria:

* Any previous diagnosis of dementia or other cognitive impairment.
* Any patient undergoing emergency surgery.
* Any patient undergoing surgery who is currently an inpatient.
* Patient refusal to participate in study.
* Any patient undergoing surgery that would prevent placement of the Sedline monitor leads (for example - surgery on the patient's forehead/scalp).
* Any physical, mental, or medical conditions which, in the opinion of the investigators, may confound the ability to assess the patient for delirium in the post-operative period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Webb, MD, Principal Investigator — Indiana University
Locations (1):
- IU Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hajat Z, Ahmad N, Andrzejowski J. The role and limitations of EEG-based depth of anaesthesia monitoring in theatres and intensive care. Anaesthesia. 2017 Jan;72 Suppl 1:38-47. doi: 10.1111/anae.13739. PMID 28044337
- [Background] MacKenzie KK, Britt-Spells AM, Sands LP, Leung JM. Processed Electroencephalogram Monitoring and Postoperative Delirium: A Systematic Review and Meta-analysis. Anesthesiology. 2018 Sep;129(3):417-427. doi: 10.1097/ALN.0000000000002323. PMID 29912008
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Wildes TS, Mickle AM, Ben Abdallah A, Maybrier HR, Oberhaus J, Budelier TP, Kronzer A, McKinnon SL, Park D, Torres BA, Graetz TJ, Emmert DA, Palanca BJ, Goswami S, Jordan K, Lin N, Fritz BA, Stevens TW, Jacobsohn E, Schmitt EM, Inouye SK, Stark S, Lenze EJ, Avidan MS; ENGAGES Research Group. Effect of Electroencephalography-Guided Anesthetic Administration on Postoperative Delirium Among Older Adults Undergoing Major Surgery: The ENGAGES Randomized Clinical Trial. JAMA. 2019 Feb 5;321(5):473-483. doi: 10.1001/jama.2018.22005. PMID 30721296
- [Background] 4. Kaplan LJ, Bailey H. Bispectral index (BIS) monitoring of ICU patients on continuous infusion of sedatives and paralytics reduces sedative drug utilization and cost.
- [Background] Ishizawa Y. Special article: general anesthetic gases and the global environment. Anesth Analg. 2011 Jan;112(1):213-7. doi: 10.1213/ANE.0b013e3181fe02c2. Epub 2010 Nov 3. PMID 21048097

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Prior to the induction of anesthesia, the Sedline monitor will be placed on the patient's head to ensure the monitor is working properly. For those in the control group, an apparatus will be placed over the monitor will not be in view of the anesthesiologist.
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 55 | 55
Completed | 51 | 51
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 51 | 51 | 102
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 30 | 31 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51 | 51 | 102
Height [Mean (Standard Deviation); unit: centimeters] | 171 (12) | 171 (11) | 171 (11)
Weight [Mean (Standard Deviation); unit: kilograms] | 80 (20) | 79 (20) | 80 (20)
BMI [Mean (Standard Deviation); unit: kilograms / meters^2] | 27 (6) | 27 (6) | 27 (6)
Baseline Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 131 (19) | 139 (22) | 135 (21)
Baseline Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 74 (12) | 80 (15) | 77 (14)
ASA physical status [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) physical status classification system is used to evaluate fitness of patients before surgery.
  1. Healthy person.
  2. Mild systemic disease.
  3. Severe systemic disease.
  4. Severe systemic disease that is a constant threat to life.
  5. A moribund person who is not expected to survive without the operation.
  Participants
    ASA 2 | 1 | 7 | 8
    ASA 3 | 49 | 43 | 92
    ASA 4 | 1 | 1 | 2
Opioid Naïve or Tolerant [Count of Participants; unit: Participants]
  Naïve | 44 | 35 | 79
  Tolerant | 7 | 16 | 23
Type of Surgery [Count of Participants; unit: Participants]
  GI/Colorectal | 33 | 31 | 64
  GYN | 2 | 0 | 2
  Other | 0 | 2 | 2
  Urologic | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Total Average Anesthetic
Description: total average percent of volatile anesthetic (sevoflurane) utilized while subjects are under anesthesia (maintenance phase).
Time Frame: 5 minutes after induction until the time which administration of neuromuscular blocker reversal drugs is given
Measure: Mean (Standard Deviation); unit: percentage of sevoflurane
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 51 | 51
percentage of sevoflurane | 1.1890 (0.2571) | 1.2906 (0.2069)

2. Secondary Outcome: Total Hypnotic Agents (Midazolam, Ketamine, Methadone, Hydromorphone)
Description: the total dosage of hypnotic agents administered while in the maintenance phase of anesthesia. These agents include: midazolam, methadone, and hydromorphone.
Time Frame: 5 minutes after induction until the time which administration of neuromuscular blocker reversal drugs is given
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 51 | 51
mg
  Midazolam | 1.29 (1.46) | 1.49 (1.46)
  Ketamine | 43.98 (38.54) | 45.40 (42.95)
  Hydromorphone | 0.39 (0.57) | 0.41 (0.47)
  Methadone | 1.18 (0.80) | 4.07 (3.31)

3. Secondary Outcome: Time Period of Hypotension
Description: this will be defined as an episode of mean arterial pressure of <65 mmHg
Time Frame: 5 minutes after induction until the time which administration of neuromuscular blocker reversal drugs is given
Measure: Mean (Standard Deviation); unit: minutes (with MAP < 65)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 51 | 51
minutes (with MAP < 65) | 27.18 (31.43) | 27.41 (34.52)

4. Secondary Outcome: Total Dosage of Vasopressor (Norepinephrine, Phenylephrine)
Description: phenylephrine, norepinephrine
Time Frame: 5 minutes after induction until the time which administration of neuromuscular blocker reversal drugs is given
Population: Please note, the units listed below are the standard units used in clinical practice for these medications
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 51 | 51
mcg
  Phenylephrine | 1442.55 (1489.29) | 4077.20 (2845.07)
  Norepinephrine | 79.45 (70.08) | 374.62 (330.02)

5. Secondary Outcome: Occurrence of EEG Isoelctricity
Description: Following the procedure, images and data from the Sedline device were evaluated to determine what percentage of the case a patient's processed EEG displayed isoelectricity (burst suppression). A burst-suppression (or suppression-burst) pattern is a discontinuous EEG, with periods of marked suppression or isoelectric intervals alternating with "bursts" of activity, with or without embedded epileptiform features (Bauer et al., 2013)
Time Frame: 5 minutes after induction until administration of neuromuscular blocker reversal drugs up to 24 hours
Measure: Mean (Standard Deviation); unit: % (of case with burst suppression)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 51 | 51
% (of case with burst suppression) | 13.60 (24.85) | 21.28 (32.58)

6. Secondary Outcome: Total Dosage of Vasopressor (Ephedrine)
Description: ephedrine
Time Frame: 5 minutes after induction until the time which administration of neuromuscular blocker reversal drugs is given
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 51 | 51
mg | 17.06 (18.26) | 13.86 (22.9)

7. Secondary Outcome: Total Dosage of Vasopressor (Vasopressin)
Description: vasopressin
Time Frame: 5 minutes after induction until the time which administration of neuromuscular blocker reversal drugs is given
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 51 | 51
Units | 0.84 (0.59) | 2.63 (1.84)

8. Secondary Outcome: Total Hypnotic Agents (Fentanyl)
Description: the total dosage of hypnotic agents administered while in the maintenance phase of anesthesia; fentanyl.
Time Frame: 5 minutes after induction until the time which administration of neuromuscular blocker reversal drugs is given
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 51 | 51
mcg | 139.22 (69.33) | 173.04 (101.22)

ADVERSE EVENTS:
Time Frame: Approx 24 hrs.
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT05051982/Prot_SAP_000.pdf